CLINICAL TRIAL: NCT04510337
Title: Does Adding Magnesium Sulphate to Low Dose Rocuronium Affects the Depth of Blockade in Cancer Patients Undergoing Direct Laryngoscope Surgical Procedures
Brief Title: Does Adding Magnesium Sulphate to Low Dose Rocuronium Affects Depth of Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Lecturer of anesthesia and pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201617031.2P
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia
MeSH Terms: interventions — Rocuronium; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard rocuronium (Active Comparator): patients received rocuronium 0.6mg/kg
  Interventions: Drug: standard rocuronium dose
- Magnesium (Experimental): patients received 100 ml saline with 50mg/kg magnesium sulphate infusion over 10 minutes
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: standard rocuronium dose — 0.6 mg/kg rocuronium during induction of anesthesia
  Other Names: standard dose rocuronium
  Arms: Standard rocuronium
Drug: Magnesium sulfate — 50 mg/kg magnesium sulphate added to 0.40 mg/kg rocuronium
  Other Names: low dose rocuronium
  Arms: Magnesium

SUMMARY:
This study aim is to compare the effect of magnesium sulphate combined with low dose rocuronium versus standard dose rocuronium

DETAILED DESCRIPTION:
Comparing the effect of magnesium sulphate combined to low dose rocuronium versus standard dose rocuronium in cancer patients undergoing direct laryngoscopy for laryngeal tumors regarding intubating conditions, intraoperative relaxation, depth of anesthesia and recovery time.

ELIGIBILITY:
Inclusion Criteria:

Patients with Laryngeal tumors

ASA I-II

Age 30-70 years

Exclusion Criteria:

Renal and or hepatic insufficiency

Neuromuscular disease

Large glottic and/or supra-glottic lesions with or without breathing difficulties

Known allergy to any of the used drug

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Onset and duration of muscle relaxant | 90 minutes
  Onset time of muscle relaxant and duration

SECONDARY OUTCOMES:
Degree of muscle relaxation | 90 minutes
  depth of blockade

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Lecturer; Mohamed A Wadod, MD, Study Director — Lecturer
Locations (1):
- National Cancer Institute, Cairo, Egypt